CLINICAL TRIAL: NCT06725498
Title: A Prospective, Single-center, Open-label Phase II Clinical Study of Intra-arterial Chemotherapy Combined with Concurrent Radiotherapy and Tislelizumab-jsgr in the Treatment of T4bNanyM0 HNSCC
Brief Title: Intra-arterial Chemotherapy Combined with Radiotherapy and Immunotherapy for HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREC2023-KY073
Record Dates: First submitted 2024-11-18; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Albumin-Bound Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RT + IAC + Anti-PD-1 antibody (Experimental): Patients must undergo Multi-Disciplinary Treatment evaluation after receiving 3 cycles of neoadjuvant therapy (Tislelizumab-jsgr combined with platinum-based chemotherapy).
  For operable patients, Radical surgery followed by adjuvant standard (chemo)radiotherapy plus Tislelizumab-jsgr (Q3W 17 cycles).
  For inoperable patients, Intra-arterial Chemotherapy concurrent with Radical radiotherapy followed by Tislelizumab-jsgr (Q3W 17 cycles).
  Interventions: Drug: Tislelizumab-jsgr; Drug: Cisplatin; Drug: Albumin-Bound Paclitaxel; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Tislelizumab-jsgr — 200mg, Q3W
Drug: Cisplatin — 60-75 mg/㎡, Q3W
Drug: Albumin-Bound Paclitaxel — 260 mg/㎡, Q3W
Radiation: Radiotherapy — Radical Radiotherapy or adjuvant Radiotherapy per guidelines.

SUMMARY:
This study pioneers a novel approach by integrating a new auxiliary chemo-immunotherapy regimen, which is then followed by an evaluation of the potential for surgical resection. For those patients who remain non-resectable, a tailored treatment plan is proposed, consisting of arterial infusion chemotherapy in conjunction with radiotherapy, succeeded by a series of immune checkpoint inhibitors. The efficacy and safety of this integrated therapeutic strategy are meticulously assessed, with the goal of enhancing survival outcomes for patients with T4bNanyM0 HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T4bNanyM0 Head and neck squamous cell carcinoma (hypopharyngeal cancer, laryngeal cancer, oropharyngeal cancer or oral cavity) with a confirmed diagnosis by histology and/or cytology;
* Expected survival ≥3 months, with adequate organ function;
* Investigators believe they can safely receive treatment with PD-1 combined with platinum and albumin-bound paclitaxel;
* Age ≥18 years;
* ECOG score of 0-1;
* Measurable disease as defined by RECIST v1.1;
* Adequate bone marrow reserve and organ function: Absolute neutrophil count (ANC) ≥1,000/microliter (mcL), platelets ≥75,000/mcL, hemoglobin ≥8g/dL, without transfusion or dependence on erythropoietin (EPO) (within 7 days after assessment);
* Renal function: Serum creatinine ≤1.5 times the upper limit of normal (ULN) OR measured or calculated creatinine clearance ≥60mL/min with creatinine levels > 1.5 times the institutional ULN. (GFR can also be used in place of creatinine or CrCl). Creatinine clearance should be calculated according to institutional standards;
* Liver function: For subjects with a total bilirubin level >1.5 ULN, serum total bilirubin ≤1.5 times ULN or direct bilirubin ≤ULN; For patients with liver metastases, aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤2.5 times ULN OR ≤5 times ULN; Albumin > 2.5 mg/dL;
* Coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN, if the subject is receiving anticoagulant therapy, PT or PTT should be within the permissible range of the anticoagulant used;
* Females should agree to use contraceptive measures (such as intrauterine device (IUD), oral contraceptives, or condoms) during the study and for 6 months after the study ends; Negative serum or urine pregnancy test within 7 days before study entry, and must be non-lactating patients; Males should agree to use contraceptive measures during the study and for 6 months after the study ends.

Exclusion Criteria:

* Patients with a history of prior immunotherapy, radiotherapy, and treatment with EGFR monoclonal antibodies;
* Patients with a history of other (including unknown primary) malignant tumors within the past 5 years;
* Patients who are intolerant to radiotherapy post-surgery;
* Patients known to be allergic to the study medication or its active ingredients, excipients;
* Patients with any unstable systemic diseases, including but not limited to: severe infections, uncontrolled diabetes, unstable angina, cerebrovascular accidents or transient ischemic attacks, myocardial infarction, congestive heart failure, serious arrhythmias requiring medication, liver, kidney, or metabolic disorders;
* Patients with potential immune deficiencies, chronic infections, including HIV, hepatitis, tuberculosis (TB), or autoimmune diseases;
* Patients with potential hematological issues, including bleeding disorders, known prior gastrointestinal bleeding requiring intervention within the past 6 months, active pulmonary embolism or deep vein thrombosis (DVT) that is unstable on anticoagulation regimens;
* A history or any evidence of active noninfectious pneumonia;
* Known active central nervous system (CNS) metastases and/or leptomeningeal disease or carcinomatous meningitis. Subjects with previously treated brain metastases may participate if they are stable (no evidence of imaging progression for at least four weeks prior to the first trial treatment and any neurological symptoms have returned to baseline), with no new or enlarging evidence of brain metastases, and are not on steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability;
* Concurrent use (or receipt) of medications within 7 days prior to Day 1 of Cycle 1 that may affect drug metabolism;
* Pregnant or breastfeeding, or expecting to become pregnant or father a child during the anticipated trial period;
* Any uncontrollable concomitant diseases, including but not limited to persistent or active infections, symptomatic congestive heart failure, unstable angina, arrhythmias;
* Prolonged corrected QT (QTc) interval > 475 ms on screening EKG;
* Ejection fraction <40% on 2D echocardiogram (ECHO) at screening;
* Any serious medical or psychiatric illness/condition, including substance use disorders, that may interfere with or limit adherence to study requirements/treatment in the investigator's judgment;
* Active autoimmune disease requiring systemic treatment in the past 2 years (i.e., the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapies (e.g., thyroid hormone, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency, etc.) are not considered a form of systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
1 year Event-free Survival rate (1y-EFS rate) | 1 year
  EFS is the time from the starting date of neoadjuvant therapy to the date of first record of any of the following events: radiographic disease progression; local or distant progression or recurrence as assessed with imaging or biopsy as indicated; or death due to any cause. Radiographic disease progression during neoadjuvant phase that precludes surgery will be considered an event; a secondary malignancy will not be considered an event.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 30 days post-neoadjuvant
  ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
Pathological Complete Response (pCR) | Up to 30 days post-surgery
  Pathological complete response (pCR) is measured as the percentage of participants with a pathological complete response as assessed by the central pathologist at the time of definitive surgery. pCR is defined as having no residual invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes.
Major Pathological Response (MPR) | Up to 30 days post-surgery
  The percentage of participants with a major pathological response (mPR) as assessed by the Central Pathologist at the time of definitive surgery. mPR is defined as ≤10% invasive squamous cell carcinoma within the resected primary tumor specimen and all the sampled regional lymph nodes.
Overall Survival (OS) | Up to 5 years
  OS was defined as the time from starting date of neoadjuvant therapy to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
Percentage of Participants Experiencing An Adverse Event (AEs) | through study completion, an average of 2 years
  Percentage of participants experiencing any sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study therapy
Local Recurrence-free Survival (LRFS) | through study completion, an average of 5 years
  Percentage of patients in a treatment group who are alive without local recurrence.
Distant Metastases-free Survival (DMFS) | through study completion, an average of 5 years
  DMFS will be defined as the time between the date of randomization and the date of first distant metastasis or date of death (whatever the cause), whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No